CLINICAL TRIAL: NCT04876664
Title: Clinical Evaluation of Continuous Non-Invasive Blood Pressure Monitors With Adult Volunteers
Brief Title: Evaluation of Continuous Non Invasive Blood Pressure With Adult Volunteers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 210080046
Record Dates: First submitted 2021-04-20; First posted 2021-05-06 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-04

CONDITIONS: Blood Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ambulatory monitoring solution (Experimental): this study has only one arm
  Interventions: Device: measuring blood pressure with noninvasive blood pressure device

INTERVENTIONS:
Device: measuring blood pressure with noninvasive blood pressure device — To measure blood pressure in different circumstances with noninvasive blood pressure device

SUMMARY:
A study to collect data recorded by devices for cNIBP evaluation purposes.

DETAILED DESCRIPTION:
The study is going to be conducted to collect data from the devices used in the study for future AMS engineering purposes as deemed appropriate by the Sponsor.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female, aged 18 years or older (≥18 years);
* Willing and able to give informed consent for participation in the study;
* Able and willing to comply with all the study requirements.

Exclusion Criteria:

* Who is pregnant or lactating;
* Who is a smoker;
* Who has consumed alcohol in the last 24 hours;
* Who has been previously diagnosed with Ataxia or balance disorder;
* Who has been previously diagnosed with Raynaud's disease/ syndrome/ phenomenon;
* Who has been previously a diagnosed cardiovascular condition requiring medication or has an internal pacemaker;
* Who has an injury, deformity, A-V fistula, or other characteristic limiting the placing of cuffs on arms/fingers;

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Data collection of NIBP measurement | through study completion, average of one day
  To collect data recorded by devices for cNIBP evaluation purposes.

SECONDARY OUTCOMES:
Collect number of adverse events (AEs), serious adverse events (SAEs), and device issues | through study completion, an average of one day
  The safety objective is to collect safety information, including type and number of adverse events (AE), serious adverse events (SAE), and device issues.

CONTACTS AND LOCATIONS:
Overall Officials: Juha Pärkkä, Principal Investigator — VTT